CLINICAL TRIAL: NCT00700180
Title: A Randomized, Open-label Study to Explore the Correlation of Biomarkers With Response Rate in Chemo-naive Patients With Advanced or Recurrent Non-squamous Non-small Cell Lung Cancer Who Receive Treatment With Avastin in Addition to Carboplatin-based Chemotherapy
Brief Title: A Study of Avastin (Bevacizumab) in Combination With Carboplatin-Based Chemotherapy in Patients With Advanced or Recurrent Non-Squamous Non-Small Cell Lung Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21015; 2008-000662-23
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Carboplatin-based chemotherapy
- 2 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: Carboplatin-based chemotherapy

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 7.5mg/kg iv on day 1 of each 3 week cycle
  Arms: 1
Drug: bevacizumab [Avastin] — 15mg/kg iv on day 1 of each 3 week cycle
  Arms: 2
Drug: Carboplatin-based chemotherapy — As prescribed

SUMMARY:
This study will explore the correlation of biomarkers with response rate, and the overall efficacy and safety, of Avastin in combination with carboplatin-based chemotherapy in patients with advanced or recurrent non-squamous non-small cell lung cancer. Patients will be randomized to one of 2 groups, to receive either Avastin 7.5mg/kg iv on day 1 of each 3 week cycle, or Avastin 15mg/kg iv on day 1 of each 3 week cycle; all patients will also receive treatment with carboplatin and either gemcitabine or paclitaxel for a maximum of 6 cycles. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* locally advanced metastatic or recurrent non-squamous non-small cell lung cancer (NSCLC);
* >=1 measurable tumor lesion;
* ECOG performance status 0-1.

Exclusion Criteria:

* prior chemotherapy or treatment with another systemic anti-cancer agent;
* evidence of CNS metastases;
* history of grade 2 or higher hemoptysis;
* evidence of tumor invading or abutting major blood vessels;
* malignancies other than NSCLC within 5 years prior to randomization, other than adequately treated cancer in situ of cervix, basal or squamous cell skin cancer, localized prostate cancer or DCIS;
* clinically significant cardiovascular disease;
* current or recent use of aspirin (>325mg/day) or full dose anticoagulants or thrombolytic agents for therapeutic purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2008-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (49):
- Australia (4):
  - St Leonards, New South Wales
  - Adelaide, South Australia
  - Box Hill, Victoria
  - Fitzroy, Victoria
- Belgium (2):
  - Antwerp
  - Liège
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario
- Czechia (2):
  - Ostrava
  - Prague
- Odense, Denmark
- France (2):
  - Paris
  - Rouen
- Germany (4):
  - Bad Berka
  - Großhansdorf
  - Hamburg
  - Oldenburg
- Hong Kong, Hong Kong
- Hungary (5):
  - Budapest
  - Edelény
  - Sopron
  - Szombathely
  - Törökbálint
- Italy (3):
  - Milan
  - Orbassano
  - Roma
- Netherlands (5):
  - Enschede
  - Hoorn
  - Nieuwegein
  - Rotterdam
  - The Hague
- Poland (3):
  - Poznan
  - Warsaw
  - Zabrze
- Russia (6):
  - Arkhangelsk
  - Chelyabinsk
  - Kazan'
  - Krasnodar
  - Moscow
  - Saint Petersburg
- Spain (3):
  - Seville, Sevilla
  - Valencia, Valencia
  - Barakaldo, Vizcaya
- Taiwan (3):
  - Changhua
  - Taichung
  - Taipei
- United Kingdom (3):
  - Aberdeen
  - Chelmsford
  - London

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab 7.5 Milligrams (mg) Plus Chemotherapy: Cycles 1-6 (3-week cycles): Participants received bevacizumab 7.5 mg per kilogram (mg/kg) intravenously (IV) on Day 1; either carboplatin at a dose required to achieve an area under the concentration-time curve (AUC) of 6 mg per milliliter (mg/mL) IV and paclitaxel 200 mg per square meter (mg/m^2) IV on Day 1, or carboplatin at AUC 5 mg/mL IV on Day 1 and gemcitabine 1200 mg/m^2 IV on Days 1 and 8. The choice of chemotherapy doublet, either carboplatin/paclitaxel or carboplatin/gemcitabine, was left to the discretion of the investigator. The cycle was repeated until disease progression or for a maximum of 6 cycles.
  Cycle 7 and beyond (3-week cycles): If the first 6 cycles were tolerated with no disease progression, participants then received bevacizumab 7.5 mg/kg IV on Day 1. This cycle was repeated every 3 weeks until disease progression.
- Bevacizumab 15 mg Plus Chemotherapy: Cycles 1-6 (3-week cycles): Participants received bevacizumab 15 mg/kg IV on Day 1; either carboplatin at a dose required to achieve an AUC of 6 mg/mL IV and paclitaxel 200 mg/m^2 IV on Day 1, or carboplatin at AUC 5 mg/mL IV on Day 1 and gemcitabine 1200 mg/m^2 IV on Days 1 and 8. The choice of chemotherapy doublet, either carboplatin/paclitaxel or carboplatin/gemcitabine, was left to the discretion of the investigator. The cycle was repeated until disease progression or for a maximum of 6 cycles.
  Cycle 7 and beyond (3-week cycles): If the first 6 cycles were tolerated with no disease progression, participants then received bevacizumab 15 mg/kg IV on Day 1. This cycle was repeated every 3 weeks until disease progression.
Period: Overall Study
Arm/Group | Bevacizumab 7.5 Milligrams (mg) Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Started | 154 | 149
Completed | 0 (Clinical cutoff date: July 11, 2011) | 0 (Clinical cutoff date: July 11, 2011)
Not Completed | 154 | 149
Not completed — Death | 99 | 114
Not completed — Alive on treatment | 5 | 3
Not completed — Alive in follow-up | 46 | 27
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population. The ITT population included all participants randomized into the study.
Groups:
- Bevacizumab 7.5 mg Plus Chemotherapy: Cycles 1-6 (3-week cycles): Participants received bevacizumab 7.5 mg/kg IV on Day 1; either carboplatin at a dose required to achieve an AUC of 6 mg/mL IV and paclitaxel 200 mg/m^2 IV on Day 1, or carboplatin at AUC 5 mg/mL IV on Day 1 and gemcitabine 1200 mg/m^2 IV on Days 1 and 8. The choice of chemotherapy doublet, either carboplatin/paclitaxel or carboplatin/gemcitabine, was left to the discretion of the investigator. The cycle was repeated until disease progression or for a maximum of 6 cycles.
  Cycle 7 and beyond (3-week cycles): If the first 6 cycles were tolerated with no disease progression, participants then received bevacizumab 7.5 mg/kg IV on Day 1. This cycle was repeated every 3 weeks until disease progression.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy | Total
Number analyzed (Participants) | 154 | 149 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (10.13) | 58.8 (11.20) | 59.2 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 98 | 94 | 192

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) by Dichotomized Baseline Plasma Marker Level
Description: Overall response was analyzed and correlated within dichotomized (low- and high-level) baseline plasma biomarker (basic fibroblast growth factor [bFGF], E-selection, intracellular adhesion molecule [ICAM], placental growth factor [PlGF], vascular endothelial growth factor A [VEGF A], vascular endothelial growth factor receptor [VEGFR]-1, and VEGFR-2) subgroups: low-level equals (=) less than or equal to (≤) median baseline level, high-level=greater than (>) median baseline level. Per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.0 CR defined as disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR defined as greater than or equal to (≥)30 percent (%) decrease under baseline of the sum of the longest diameter (LD) of all target lesions. No unequivocal progression of non-target disease; no new lesions. Complete and partial responses must have been confirmed no less than 4 weeks after criteria for response were first met
Time Frame: Baseline, Day 21 of Cycles 2, 4, and 6 (Bv + chemo), Day 21 of Cycles 7, 8, 9, and 10 (Bv), Day 21 of every other cycle (Bv), and at disease progression.
Population: Biomarker Evaluable Protein Plasma (BEP) Population: Participants in the ITT population who started at least 1 dose of bevacizumab and had a non-missing baseline biomarker level determined for at least 1 biomarker. n (number) equals (=) number of participants assessed for the specified biomarker.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 82 | 75
percentage of participants
  bFGF low level (n=77,65) | 42.86 | 47.69
  bFGF high level (n=66,75) | 34.85 | 49.33
  E-selectin low level (n=73,69) | 36.99 | 42.03
  E-selectin high level (n=70,71) | 41.43 | 54.93
  ICAM low level (n=70,72) | 38.57 | 50.00
  ICAM high level (n=29,32 | 39.73 | 47.06
  PlGF low level (n=82, 64) | 37.80 | 51.56
  PlGF high level (n=27,29) | 33.33 | 51.72
  VEGF A low level (n=73,67) | 42.47 | 44.78
  VEGF A high level (n=67,73) | 35.82 | 53.42
  VEGFR-1 low level (n=72,70) | 37.50 | 60.00
  VEGFR-1 high level (n=71,70) | 40.85 | 37.14
  VEGFR-2 low level (n=74,69) | 32.43 | 46.38
  VEGFR-2 high level (n=69,71) | 46.38 | 50.70
Statistical Analysis 1: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy; bFGF (high versus low); Test type: Superiority or Other; p = 0.8127, Regression, Logistic — Multiple logistic regression model with treatment, biomarker level (dichotomized) and baseline prognostic factors as covariates; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.63 to 1.80]
Statistical Analysis 2: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy; E-selectin (high versus low); Test type: Superiority or Other; p = 0.0285, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.06 to 3.08]
Statistical Analysis 3: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy; ICAM (high versus low); Test type: Superiority or Other; p = 0.7478, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.64 to 1.85]
Statistical Analysis 4: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy; PlGF (high versus low); Test type: Superiority or Other; p = 0.6761, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.58 to 2.33]
Statistical Analysis 5: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy; VEGF A (high versus low); Test type: Superiority or Other; p = 0.4601, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.22, 95% CI 2-sided [0.72 to 2.09]
Statistical Analysis 6: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy; VEGFR-1 (high versus low); Test type: Superiority or Other; p = 0.3193, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.77, 95% CI 2-sided [0.46 to 1.29]
Statistical Analysis 7: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy; VEGFR-2 (high versus low); Test type: Superiority or Other; p = 0.1758, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.44, 95% CI 2-sided [0.85 to 2.45]

2. Secondary Outcome: Progression-Free Survival - Percentage of Participants With an Event
Description: PFS was defined as the time between randomization and progressive disease (PD) according to RECIST criteria, or death due to any cause. PD was defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started. Disease progression was evaluated according to the RECIST using computed tomography (CT) scans, magnetic resonance imaging (MRI) scans, X-ray, bone scans, or clinical examination. Participants without an event were censored at the date of last follow up for progression. Participants with no post baseline follow-up for progression were censored at the day of randomization.
Time Frame: Baseline, Day 1, weekly to disease progression
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 154 | 149
percentage of participants | 83.1 | 85.9

3. Secondary Outcome: Progression-Free Survival - Time to Event
Description: PFS was defined as the time between randomization and disease progression or death due to any cause. Participants without an event were censored at the date of last follow up for progression. Participants with no post baseline follow-up for progression were censored at the day of randomization. Disease progression was evaluated according to the RECIST using CT scans, MRI scans, X-ray, bone scans, or clinical examination. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Baseline, Day 1, weekly to disease progression
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 154 | 149
months | 6.8 [5.9 to 7.4] | 6.7 [5.9 to 7.2]
Statistical Analysis 1: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy vs Bevacizumab 15 mg Plus Chemotherapy; Test type: Superiority or Other; p = 0.9454, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.78 to 1.31]

4. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with CR or PR according to RECIST criteria. Per RECIST v1.0: CR defined as disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR was defined as ≥30% decrease under baseline of the sum of the LD of all target lesions. No unequivocal progression of non-target disease. No new lesions. Complete and partial responses were confirmed no less than 4 weeks after the criteria for response were first met.
Time Frame: Baseline, Day 21 of Cycles 2, 4, and 6, Day 21 of Cycles 7, 8, 9, and 10, Day 21 of every other cycle, and at disease progression
Population: ITT Population. Data for 12 participants (3 at 7.5 mg and 9 at 15 mg) were excluded for reasons including but not limited to: no study treatment (ST), no postbaseline tumor assessment (TA), non-protocol defined antineoplastic therapy before first TA, first TA >70 days after last dose of last ST, last TA less than (<) 42 days from start of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 154 | 149
percentage of participants | 37.1 [29.4 to 45.3] | 46.4 [38.0 to 55.0]
Statistical Analysis 1: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy vs Bevacizumab 15 mg Plus Chemotherapy; Test type: Superiority or Other; p = 0.1737, Cochran-Mantel-Haenszel; Difference in Responses Rates = 9.34, 95% CI 2-sided [-2.4 to 21.0] — Approximate 95% Confidence Interval (CI) for difference of two rates using Hauck-Anderson method

5. Secondary Outcome: Percentage of Participants With Measurable Disease at Baseline Who Achieved CR, PR, or Stable Disease (SD) for at Least 6 Weeks
Description: Percentage of participants with measurable disease at baseline who on assessment achieved CR, PR, or SD according to RECIST. Per RECIST v1.0: CR defined as disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR was defined as ≥30% decrease under baseline of the sum of the LD of all target lesions. No unequivocal progression of non-target disease. No new lesions. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since start of treatment. Complete and partial responses must have been confirmed no less than 4 weeks after the criteria for response were first met. For participants with SD, follow-up assessments must have met the SD criteria at least once after study entry at a minimum interval of 6 weeks.
Time Frame: as for outcome 4
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 151 | 140
percentage of participants | 76.8 [69.3 to 83.3] | 78.6 [70.8 to 85.1]
Statistical Analysis 1: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy vs Bevacizumab 15 mg Plus Chemotherapy; Test type: Superiority or Other; p = 0.6148, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 1.75, 95% CI 2-sided [-8.2 to 11.7] — Approximate 95% CI for difference of two rates using Hauck-Anderson method

6. Secondary Outcome: Duration of Response - Percentage of Participants With an Event
Description: Duration of response is defined as time in months from the first documentation of objective tumor response (CR or PR) to objective tumor progression or death due to any cause. Participants without an event (documented progression or death) were censored at the date of last follow-up for progression. Duration of response was only calculated for participants who had a confirmed objective tumor response (CR or PR).
Time Frame: as for outcome 4
Population: ITT population; only participants with an objective tumor response (CR or PR) were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 56 | 65
percentage of participants | 80.4 | 78.5

7. Secondary Outcome: Duration of Response - Time to Event
Description: The median time, in months, from the first documentation of objective tumor response (CR or PR) to objective tumor progression or death due to any cause. Participants without an event (documented progression or death) were censored at the date of last follow-up for progression. Duration of response was only calculated for participants who had a confirmed objective tumor response (CR or PR). Median Duration of Response was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: ITT population: only participants with an objective tumor response (CR or PR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 56 | 65
months | 5.8 [5.2 to 7.0] | 5.6 [4.6 to 7.1]
Statistical Analysis 1: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy vs Bevacizumab 15 mg Plus Chemotherapy; Test type: Superiority or Other; p = 0.7587, Log Rank; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.68 to 1.69]

8. Secondary Outcome: Overall Survival - Percentage of Participants With an Event
Description: Overall survival was defined as the time between randomization and death due to any cause. Participants without an event were censored at the last time they were known to be alive. Overall Survival was estimated using the Kaplan-Meier method.
Time Frame: Baseline, weekly to 28 days after last dose of study treatment, every 8 weeks thereafter to death due to any cause
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 154 | 149
percentage of participants | 64.3 | 76.5

9. Secondary Outcome: Overall Survival - Time to Event
Description: as for outcome 8
Time Frame: Baseline, weekly to death due to any cause, or to end of study
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Number analyzed (Participants) | 154 | 149
months | 13.4 [10.5 to 18.1] | 13.7 [11.4 to 17.0]
Statistical Analysis 1: Comparison: Bevacizumab 7.5 mg Plus Chemotherapy vs Bevacizumab 15 mg Plus Chemotherapy; Test type: Superiority or Other; p = 0.3120, Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.87 to 1.53]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from first study treatment until 28 days after last study treatment (LST). In addition, surgical procedures, major injuries and adverse events of special interest for bevacizumab were assessed to at least 6 months after LST.
Arm/Group | Bevacizumab 7.5 mg Plus Chemotherapy | Bevacizumab 15 mg Plus Chemotherapy
Serious Adverse Events (participants affected / at risk) | 53/151 | 57/143
Other Adverse Events (participants affected / at risk) | 137/151 | 132/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 7.5 mg Plus Chemotherapy (N=151) | Bevacizumab 15 mg Plus Chemotherapy (N=143)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 13
Neutropenia (Blood and lymphatic system disorders) | 13 | 7
Anaemia (Blood and lymphatic system disorders) | 10 | 8
Granulocytopenia (Blood and lymphatic system disorders) | 3 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Bone Marrow Failure (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Artery Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 5 | 7
Pyothorax (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Localised Infection (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 0 | 1
Pneumonia Legionella (Infections and infestations) | 0 | 1
Pseudomonal Sepsis (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 1 | 5
Death (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Cerebral Infarction (Nervous system disorders) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 1
Embolic Stroke (Nervous system disorders) | 0 | 1
Ischaemic Stoke (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 0 | 2
Myocardial Infarction (Cardiac disorders) | 2 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Palapitations (Cardiac disorders) | 1 | 0
Tachycardia Paroxysmal (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Intestinal Perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypertensive Crisis (Vascular disorders) | 1 | 1
Arterial Thrombosis (Vascular disorders) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Intestinal Anastomosis Complication (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Fluid Retension (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Renal Scan Abnormal (Investigations) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab 7.5 mg Plus Chemotherapy (N=151) | Bevacizumab 15 mg Plus Chemotherapy (N=143)
Neutropenia (Blood and lymphatic system disorders) | 72 | 57
Thrombocytopenia (Blood and lymphatic system disorders) | 62 | 41
Anaemia (Blood and lymphatic system disorders) | 54 | 39
Leukopenia (Blood and lymphatic system disorders) | 28 | 16
Nausea (Gastrointestinal disorders) | 52 | 38
Constipation (Gastrointestinal disorders) | 27 | 20
Vomiting (Gastrointestinal disorders) | 18 | 22
Diarrhoea (Gastrointestinal disorders) | 19 | 16
Stomatitis (Gastrointestinal disorders) | 9 | 9
Mouth ulceration (Gastrointestinal disorders) | 12 | 5
Abdominal pain upper (Gastrointestinal disorders) | 10 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 33 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 22
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Fatigue (General disorders) | 47 | 41
Chest pain (General disorders) | 19 | 9
Pyrexia (General disorders) | 17 | 7
Asthenia (General disorders) | 13 | 10
Mucosal inflammation (General disorders) | 10 | 9
Dizziness (Nervous system disorders) | 17 | 16
Neuropathy peripheral (Nervous system disorders) | 19 | 10
Headache (Nervous system disorders) | 16 | 12
Dysgeusia (Nervous system disorders) | 10 | 8
Polyneuropathy (Nervous system disorders) | 5 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 35 | 30
Rash (Skin and subcutaneous tissue disorders) | 15 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 7
Hypertension (Vascular disorders) | 27 | 30
Decreased appetite (Metabolism and nutrition disorders) | 16 | 26
Weight decreased (Investigations) | 14 | 13
Alanine aminotransferase increased (Investigations) | 9 | 4
Nasopharyngitis (Infections and infestations) | 14 | 13
Urinary tract infection (Infections and infestations) | 8 | 8
Proteinuria (Renal and urinary disorders) | 12 | 17
Insomnia (Psychiatric disorders) | 12 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.